CLINICAL TRIAL: NCT03024437
Title: A Phase I/II Study to Evaluate the Safety, Pharmacodynamics and Efficacy of Atezolizumab in Combination With Entinostat and Bevacizumab in Patients With Advanced Renal Cell Carcinoma
Brief Title: Atezolizumab in Combination With Entinostat and Bevacizumab in Patients With Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Genentech has closed the study due to lack of data with Atezo
Sponsor: Roberto Pili (Other)
Collaborators: Genentech, Inc. (Industry); Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Roberto Pili, Professor of Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0574
Record Dates: First submitted 2017-01-16; First posted 2017-01-18 (Estimated); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Cancer; Renal Cancer
Keywords: PD-L1 inhibitor
MeSH Terms: conditions — Neoplasm Metastasis; Kidney Neoplasms | interventions — atezolizumab; Bevacizumab; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Dose Escalation (Experimental): Open to patients meeting eligibility criteria with advanced renal cell carcinoma and ANY or NO prior treatments.
  Three dose levels of entinostat will be tested in 3-patient cohorts according to the 3 + 3 standard design (1 mg, 3 mg and 5 mg). The starting dose level of entinostat will be 1 mg orally every 7 days. The Phase II dose will be recommended phase II dose of entinostat (i.e., the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor).
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Entinostat
- Phase II - Cohort A (Experimental): Open to patients meeting eligibility criteria with advanced renal cell carcinoma and NO prior treatments.
  Patients in Cohort A will be treated with atezolizumab, bevaciuzmab, and the recommended phase II dose of entinostat. During Phase II, the study will have a run-in period with entinostat for one cycle followed by atezolizumab and bevacizumab for the second cycle, and then the combination phase (i.e., atezolizumab + bevacizumab + entinostat for all cycles thereafter).
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Entinostat
- Phase II - Cohort B (Experimental): Open to patients meeting eligibility criteria with advanced renal cell carcinoma and at least one prior treatment with a PD1 or PDL1 inhibitor.
  Patients in Cohort B will be treated with the same combination therapy as in Cohort A.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Entinostat

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be given intravenously every 3 weeks at 1200 mg.
  Other Names: MDPL3280A
Drug: Bevacizumab — Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg.
  Other Names: Avastin
Drug: Entinostat — Entinostat will be given orally every 7 days at 1, 3, or 5 mg depending upon phase. In Phase I, dose levels will be tested in up to 3 cohorts starting at 1 mg. In Phase II, the dose will be the recommended phase II dose that was determined during Phase I (i.e., 1, 3, or 5 mg).
  Other Names: SNDX-275

SUMMARY:
This study will assess the immunomodulatory activity of entinostat in patients with advanced renal cell carcinoma receiving the PD-L1 inhibitor atezolizumab. The overall hypothesis is that entinostat will increase the immune response and anti-tumor effect induced by the PD-L1 inhibition by suppressing Treg function. We have chosen renal cell carcinoma that has been reported to respond to PD1/PD-L 1 inhibition. The schedule of entinostat is based on our previous experience with this agent. Based on our working hypothesis that low dose HDAC inhibitors will have a suppressive function on Tregs but not on T effector cells, the starting dose of entinostat will be 1 mg and will be escalated up to 5 mg rather than the 10 mg dose. The combination also with bevacizumab will provide an effective VEGF inhibition that may potentiate the immune response and anti-tumor effect induced by atezolizumab. The proposed dose and schedule for atezolizumab and bevacizumab has been shown to be well tolerated in prior Phase/I/II studies and is currently tested in a Phase III randomized study in patients with renal cell carcinoma with sunitinib as a control arm. The highest proposed dose level for entinostat (5 mg) represents 50% of the recommended Phase II dose for this compound as a single agent.

DETAILED DESCRIPTION:
This is a Phase l/II, open-label, safety, pharmacodynamics and efficacy study of atezolizumab in combination with entinostat and bevacizumab in patients with advanced renal cell carcinoma. This clinical study will be composed of a Dose Finding Phase (Phase I) and a two-stage Phase (Phase II) portion.

In Phase 1 Combination Phase), patients will be treated with oral entinostat every 7 days, with bevacizumab at the fixed dose of 15 mg/kg IV every 3 weeks and with atezolizumab at the fixed dose of 1200 mg IV every 3 weeks. Each cycle length is 21 days. Three dose levels of entinostat will be tested in 3-design patient cohorts according to the 3 + 3 standard design (1 mg, 3 mg and 5 mg). For the Dose Finding Phase, the starting dose level of pill be 1 mg by mouth every 7 days. The first dose level will have a minimum of 3 patients treated (unless the first 2 patients experience DLT(s) before the 3rd patient is enrolled). DLTs attributable to entinostat and/or bevacizumab and/or atezolizumab will be evaluated during the first 21 days of the combination treatment.

If a DLT occurs in 1 patient treated at the starting dose level, a minimum of 3 additional patients will be treated at this dose level. If DLTs occur in 2 or more of the first 6 patients, the study will be terminated. If a DLT occurs in 1 out of 6 patients, 3 additional patients will be treated at the next dose level (level 2). If no DLTs occur at the starting dose level 1, 3 additional patients will be treated at the next dose level (level 2). If no DLTs occur at the dose level 2, 3 additional patients will be treated at the next dose level (level 3). If no DLTs occur at dose level 3, this dose level will be recommended for the Phase II portion of the study. Patients who experience Grade ≥ 3 toxicity and recover to ≤ Grade 1 (or to pretreatment baseline level toxicity) may continue treatment at the next lower level. The Phase II Dose will be RP2D of entinostat (i.e., the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor-Investigator).

Once the RP2D is identified, the Phase II portion (Simon's two stage design) will be opened. During Phase II, Cohorts A and B will have a Run-In period with entinostat for one cycle followed by atezolizumab and bevacizumab for the second cycle, and then the Combination Phase. The reason for the Run-In period is to obtain data on the immunomodulatory effects of entinostat separately from bevacizumab and atezolizumab. The run-in period will be optional for patients, including those who are rapidly progressing, or if it is in the patient's best interest clinically as determined by the treating physician's discretion. In Stage I, 27 patients with prior treatments will be enrolled in two Phase II cohorts: 18 treatment naïve (anti-PD1/PDL1 naïve) patients (Cohort A), and 9 anti-PD1 resistant (defined as patients who have been on PD1 inhibitors for at least 3 months and have progressed by either clinical or radiographic assessment) patients (Cohort B). If ≥ 5 responses are observed and confirmed in Cohort A, Stage II will be conducted with 15 additional patients. In Cohort B, if any patients has a response that is observed and confirmed, Stage II will be conducted with 7 additional patients. Patients will be treated on Cohort B with the same combination therapy as in Cohort A.

Cohort B is a pilot arm which aims to test atezolizumab in anti-PD1 resistant patients. If there is no response to atezolizumab, then the RP2D dose of entinostat will be added to the standard dose of atezolizumab. If there is a response to atezolizumab, patients will continue to be treated with atezolizumab alone.

The RP2D is the dose of entinostat, atezolizumab, and bevacizumab in combination chosen for further clinical development. Further experience in the Dose Expansion Cohort may result in a RP2D dose lower than the MTD.

Objectives:

1. Primary Phase I: To assess the safety and tolerability of atezolizumab in combination with entinostat and bevacizumab in patients with advanced renal cell carcinoma.
2. Primary Phase II: To assess the objective response rate of atezolizumab in combination with entinostat and bevacizumab in anti-PD 1 naïve patients and atezolizumab in combination with entinostat in anti-PD 1 resistant patients with advanced renal cell carcinoma.
3. Secondary: To assess the objective response rate (Phase I only), progression-free survival and overall survival.
4. Correlative: To characterize PD-L1/2, immune cell subsets, and miRs in tumor and/or blood in correlation with response.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

* Signed Informed Consent Form (ICF)
* Ability and willingness to comply with the requirements of the study protocol
* Age ≥ 18 years
* Measurable disease per RECIST v1.1 (see Appendix 4) for patients with solid malignancies or patients with bone disease must have disease evaluable by bone scan and/or PET scan
* Metastatic renal cell carcinoma

  o During Phase I - All prior treatments or none are allowed
  * During Phase II/Cohort A - No prior treatments with PD1 or PDL1 inhibitors allowed
  * During Phase II/Cohort B - Must have at least one prior treatment with a PD1 or PDL1 inhibitor for metastatic disease for at least 3 months and have progressed by either clinical or radiographic assessment
* Life expectancy of at least 6 months
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1):

  * Absolute neutrophil count (ANC) ≥ 1500 cells/microL
  * White blood cell (WBC) counts > 2500/microL
  * Lymphocyte count ≥ 300/microL
  * Platelet count ≥ 100,000/microL; for patients with hematologic malignancies, platelet count ≥ 75,000/microL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception:

Patients with known Gilbert disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.

Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN

- Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN with the following exception: Patients with liver involvement: AST and/or ALT ≤ 5 x ULN

- Alkaline phosphatase (ALP) ≤ 2.0 x ULN with the following exception: Patients with documented liver involvement or bone metastases: ALP ≤ 5 x ULN

* Serum creatinine ≤ 1.25 x ULN or creatinine clearance ≥ 60 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate estimation:

  (140 - age) x (weight in kg) x (0.85 if female) / 72 x (serum creatinine in mg/dL)
* Urine dipstick for proteinuria < 2+ or 24-hour urine protein < 1 g of protein is demonstrated
* International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation (such as low-molecular-weight heparin or warfarin) should be on a stable dose.

  • If a female of childbearing potential, negative serum blood pregnancy test during screening and a negative urine pregnancy test ≤ 3 days prior to receiving the first dose of study drug. If the screening serum test is done ≤ 3 days prior to receiving the first dose of study drug, a urine test is not required.
* Non-childbearing potential is defined as (by other than medical reasons):

  * ≥ 45 years of age and has not had menses for > 2 years
  * Amenorrheic for < 2 years without a hysterectomy and/or oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
  * Post hysterectomy or oophorectomy. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound.
  * For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use two forms of highly effective contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 150 days after the last dose of all study drugs (atezolizumab, entinostat, and bevacizumab).
  * Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria Patients who meet any of the following criteria will be excluded from study entry.

General Exclusion Criteria:

* Any approved anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, ≤ 3 weeks prior to first dose of study drug; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anti-cancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
  * Palliative radiotherapy for bone metastases > 2 weeks prior to Cycle 1, Day 1
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device ≤ 4 weeks of the first dose of study drug.
* AEs from prior anti-cancer therapy that have not resolved to Grade ≤ 1 except for alopecia and neuropathy
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
* Bisphosphonate therapy for symptomatic hypercalcemia

  * Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Patients with acute leukemias, accelerated/blast phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases - Patients with asymptomatic untreated CNS disease may be enrolled, provided all of the following criteria are met: Evaluable or measurable disease outside the CNS No metastases to brain stem, midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm) No history of intracranial hemorrhage or spinal cord hemorrhage No ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted.

No neurosurgical resection or brain biopsy ≤ 28 days prior to Cycle 1, Day 1

- Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following: Radiographic demonstration of improvement upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study No stereotactic radiation or whole-brain radiation ≤ 28 days prior to Cycle 1, Day 1 Screening CNS radiographic study ≥ 4 weeks from completion of radiotherapy and ≥ 2 weeks from discontinuation of corticosteroids

* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Known hypersensitivity to any component of bevacizumab
* Allergy to benzamide or inactive components of entinostat
* Inability to comply with study and follow-up procedures
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg) that persists over 3 weeks and 3 consecutive measurements (each one week apart) despite medication
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Uncontrolled diabetes mellitus
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible.
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

Rash must cover less than 10% of body surface area (BSA) Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%) No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)

* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  - History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* History of HIV infection (HIV 1/2 antibodies) or active hepatitis B (chronic or acute) or hepatitis C infection

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. HBV DNA test must be performed in these patients prior to study treatment.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Active tuberculosis
* Clinically significant (i.e. active) cardiovascular disease (e.g., myocardial infarction or arterial thromboembolic events ≤ 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, Grade II or greater congestive heart failure, or serious cardiac arrhythmia (see Appendix 5), or a QTc interval > 470 msec.)
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis ≤ 6 months of study enrollment
* Any previous venous thromboembolism > NCI CTCAE Grade 3
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) ≤ 28 days of study enrollment
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Current or recent (≤ 10 days of study enrollment) use of aspirin (> 325 mg/day), clopidogrel (>75 mg/day), or therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to medical standard of the institution) and the patient has been on a stable dose of anticoagulants for at least 2 week at the time of study enrollment. Prophylactic use of anticoagulants is allowed.
* Severe infections ≤ 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection ≤ 2 weeks prior to Cycle 1, Day 1
* Received oral or IV antibiotics ≤ 2 weeks prior to Cycle 1, Day 1

  - Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Major surgical procedure ≤ 28 days prior to Cycle 1, Day 1 or anticipation of need for a major pre-planned surgical procedure during the course of the study
* Administration of a live, attenuated vaccine ≤ 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study

  - Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist ®) ≤ 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* History of abdominal fistula or gastrointestinal perforation ≤ 6 months before Cycle 1, Day 1. Serious non-healing wound, active ulcer, or untreated bone fracture (adjuvant trials: bone fractures must be healed)
* Proteinuria as demonstrated by a UPC ratio ≥ 1.0 at screening
* Malignancies other than the disease under study ≤ 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] ≤ 10 mg/mL, etc.)

Medication-Related Exclusion Criteria:

* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]- α or interleukin [IL]-2) ≤ 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Treatment with investigational agent ≤ 4 weeks prior to Cycle 1, Day 1 (or within five half lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) ≤ 2 weeks prior to Cycle 1, Day 1

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Adra, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Dose Level 1: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and ANY or NO prior treatments.
  Patients in Phase I Dose Level 1 will be treated with atezolizumab, bevaciuzmab, and entinostat at a dose of 1 mg.
  Atezolizumab will be given intravenously every 3 weeks at 1200 mg. Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg. Entinostat will be given orally every 7 days at 1 mg.
- Phase I - Dose Level 2: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and ANY or NO prior treatments.
  Patients in Phase I Dose Level 2 will be treated with atezolizumab, bevaciuzmab, and entinostat at a dose of 3 mg.
  Atezolizumab will be given intravenously every 3 weeks at 1200 mg. Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg. Entinostat will be given orally every 7 days at 3 mg.
- Phase I - Dose Level 3: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and ANY or NO prior treatments.
  Patients in Phase I Dose Level 3 will be treated with atezolizumab, bevaciuzmab, and entinostat at a dose of 5 mg.
  Atezolizumab will be given intravenously every 3 weeks at 1200 mg. Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg. Entinostat will be given orally every 7 days at 5 mg.
- Phase II - Cohort A: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and NO prior treatments.
  Patients in Cohort A will be treated with atezolizumab, bevaciuzmab, and the recommended phase II dose of 5 mg of entinostat.
  Atezolizumab will be given intravenously every 3 weeks at 1200 mg. Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg. Entinostat will be given orally every 7 days at 5 mg.
- Phase II - Cohort B: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and at least one prior treatment with a PD1 or PDL1 inhibitor.
  Patients in Cohort B will be treated with atezolizumab, bevaciuzmab, and the recommended phase II dose of 5 mg of entinostat.
  Atezolizumab will be given intravenously every 3 weeks at 1200 mg. Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg. Entinostat will be given orally every 7 days at 5 mg.
Period: Overall Study
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase II - Cohort A | Phase II - Cohort B
Started | 6 | 6 | 6 | 12 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 12 | 1
Not completed — Adverse Event | 0 | 1 | 3 | 5 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0
Not completed — Disease progression, relapse | 1 | 0 | 0 | 3 | 0
Not completed — Disease progression, refractory disease | 4 | 4 | 2 | 2 | 1
Not completed — Newly diagnosed cancer | 0 | 0 | 0 | 1 | 0
Not completed — Moved out of state | 0 | 1 | 0 | 0 | 0
Not completed — Needed an alternative therapy prohibited by protocol | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase II - Cohort A | Phase II - Cohort B | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 1 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 3 | 8 | 1 | 23
  >=65 years | 0 | 1 | 3 | 4 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (9.0) | 56.8 (8.9) | 63.1 (12.0) | 59.4 (9.9) | 54.1 (NA) — Standard deviation is not applicable with a sample size of one. | 57.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 0 | 7
  Male | 5 | 4 | 4 | 10 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 5 | 11 | 1 | 28
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 5 | 11 | 0 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 12 | 1 | 31
ECOG Performance Status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. - Dead
  Participants
    0 | 3 | 3 | 5 | 9 | 1 | 21
    1 | 3 | 3 | 1 | 3 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Recommended Phase II Dose of Entinostat
Description: Three dose levels of entinostat (1 mg, 3 mg and 5 mg) were tested according to the 3 + 3 standard design. The starting dose level of entinostat was 1 mg orally every 7 days. DLTs attributable to entinostat and/or bevacizumab and/or atezolizumab were evaluated during the first 21 days of the combination treatment.
  If a DLT occurs in 1 patient treated at the starting dose level, a minimum of 3 additional patients will be treated at this dose level. If DLTs occur in 2 or more of the first 6 patients, the study will be terminated. If a DLT occurs in 1 out of 6 patients, 3 additional patients will be treated at the next dose level (level 2). If no DLTs occur at the starting dose level 1, 3 additional patients will be treated at the next dose level (level 2). The process is repeated for dose level 2. If no DLTs occur at dose level 3 or if 1 DLT occurs out of 6 patients, then this dose level will be recommended for the Phase II portion of the study.
Time Frame: 21 days
Population: Patients who received at least one cycle of study drugs and had at least one post-baseline evaluation.
Measure: Number; unit: mg
Groups:
- Phase I - Dose Escalation: Open to patients meeting eligibility criteria with advanced renal cell carcinoma and ANY or NO prior treatments.
  Three dose levels of entinostat will be tested in 3-patient cohorts according to the 3 + 3 standard design (1 mg, 3 mg and 5 mg). The starting dose level of entinostat will be 1 mg orally every 7 days.
  Atezolizumab: Atezolizumab will be given intravenously every 3 weeks at 1200 mg.
  Bevacizumab: Bevacizumab will be given intravenously every 3 weeks at 15 mg/kg.
  Entinostat: Entinostat will be given orally every 7 days at 1, 3, or 5 mg depending upon dose escalation cohort. In Phase I, dose levels will be tested in up to 3 cohorts starting at 1 mg.
Arm/Group | Phase I - Dose Escalation
Number analyzed (Participants) | 18
mg | 5

2. Primary Outcome: Phase II: Percentage of Patients With Objective Response
Description: Percentage of patients who achieved a complete response or partial response to treatment as measured per RECIST 1.1.
  Complete response: Disappearance of all target lesions. Partial response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Up to 1 year
Population: Patients who received at least one cycle of study drugs and had at least one post-baseline evaluation. Patients who were treated at Dose Level 3 in Phase I were assigned to the applicable Phase II cohort for efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II - Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 16 | 3
percentage of participants | 62.5 [35.4 to 84.8] | 33.3 [0.8 to 90.6]

3. Secondary Outcome: Phase I: Percentage of Patients With Objective Response
Description: as for outcome 2
Time Frame: Up to 1 year
Population: Patients who received at least one cycle of study drugs and had at least one post-baseline evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 6 | 5 | 6
percentage of patients | 50 [11.8 to 88.2] | 20 [0.5 to 71.6] | 83.3 [35.9 to 99.6]

4. Secondary Outcome: Phase II: Median Progression-free Survival
Description: Progression free survival was defined as the time from on treatment date to date of recurrence of any type or death from any cause. Patients who did not experience recurrence or death were censored at their last evaluation date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 4.5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II - Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 16 | 3
months | 13.7 [8.7 to 21.3] | 9.8 [1.3 to NA] — The upper limit of the 95% confidence interval could not be estimated due to an insufficient number of participants with events.

5. Secondary Outcome: Phase II: Median Overall Survival
Description: Overall survival was defined as the time from on treatment date to death due to any cause. Patients who remained alive were censored at their last known alive date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 5.5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II - Cohort A | Phase II - Cohort B
Number analyzed (Participants) | 16 | 3
months | 51.6 [21.8 to NA] — The upper limit of the 95% confidence interval could not be estimated due to an insufficient number of participants with events. | 31.2 [22.8 to NA] — The upper limit of the 95% confidence interval could not be estimated due to an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to 2.5 years for adverse events and up to 5.5 years for all-cause mortality.
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase II - Cohort A | Phase II - Cohort B
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 4/6 | 4/12 | 1/1
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 6/6 | 6/12 | 0/1
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 12/12 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=6) | Phase I - Dose Level 2 (N=6) | Phase I - Dose Level 3 (N=6) | Phase II - Cohort A (N=12) | Phase II - Cohort B (N=1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=6) | Phase I - Dose Level 2 (N=6) | Phase I - Dose Level 3 (N=6) | Phase II - Cohort A (N=12) | Phase II - Cohort B (N=1)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 1 (3) | 5 (5) | 10 (25) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (4) | 4 (5) | 3 (4) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (5) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 6 (10) | 5 (7) | 6 (11) | 0 (0)
Fever (General disorders) | 1 (2) | 2 (2) | 3 (5) | 3 (3) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (7) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (4) | 4 (8) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (6) | 1 (3) | 4 (12) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 10 (19) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Weight loss (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (4) | 1 (2) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 4 (6) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (7) | 4 (6) | 4 (5) | 9 (19) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (5) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 8 (11) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (4) | 1 (2) | 2 (2) | 9 (13) | 0 (0)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (8) | 1 (4)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT03024437/Prot_SAP_000.pdf